CLINICAL TRIAL: NCT07010289
Title: NOURISH: Nurturing Outreach for Understanding and Reducing Inpatient Security of Health
Brief Title: Nurturing Outreach for Understanding and Reducing Inpatient Security of Health
Acronym: NOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00131272
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-05

CONDITIONS: Food Insecurity
Keywords: vulnerable populations; hospitalized children; health inequity
MeSH Terms: interventions — Fast Foods; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prepared Meals (Experimental): Weekly home meal delivery for four weeks.
  Interventions: Other: Prepared Meals
- Grocery Gift Cards (Experimental): Weekly grocery store gift cards for four weeks.
  Interventions: Other: Grocery Gift Cards
- Standard of Care (Active Comparator): Provision of printed and electronic food access resources.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Prepared Meals — Participants will receive the intervention of weekly home meal delivery, consecutively for 4 weeks, delivered to their home. The meals will be provided by Providence Community Kitchen, which is a program of Second Harvest Food Bank of Northwest NC. During the 4 weeks of meal provisions, participants will receive 7 family style frozen dinners delivered to the participant's home weekly. Meals are frozen, have minimal preparation time, and can be heated by oven.
  Arms: Prepared Meals
Other: Grocery Gift Cards — Participants will receive weekly grocery store gift cards, consecutively for 4 weeks. During the 4 weeks of gift card provisions, participants will receive (1) $40.00 grocery store gift card weekly, mailed to participants' home address by study staff.
  Arms: Grocery Gift Cards
Other: Standard of Care — Participants will receive the current standard for care for families endorsing inpatient food insecurity during a hospitalization, which include provision of printed and electronic food access resources. Currently, all families with positive food insecurity screening are met by a community health worker in the hospital who reviews current food access status with families (including enrollment in federal nutrition programs) and provides them with printed and electronic resources of nearby food pantries and other food access resources available to them at time of discharge from the hospital.
  Arms: Standard of Care

SUMMARY:
Food insecurity is the lack of consistent access to the food needed for a healthy life. Food insecurity among families whose child has been hospitalized is a critical problem affecting a large, vulnerable population. The purpose of this study is to identity the most effective ways to help those families with food insecurity.

DETAILED DESCRIPTION:
To address food insecurity among families who child has been hospitalized, study objectives are 1) to demonstrate the feasibility and acceptability of providing family meals and grocery store gift cards to address food insecurity among children discharged from the hospital, and 2) evaluate the potential impact of the interventions on household food insecurity, 30-day readmission rates, and primary care follow up. To accomplish these objectives, this pilot feasibility trial will be conducted at Atrium Health Levine Children's-Brenner Children's Hospital, an academic medical center that serves communities with high rates of food insecurity, in collaboration with our long-term partner Second Harvest Food Bank of Northwest North Carolina. The will recruit families whose child was admitted to the hospital and screened positive for food insecurity. All families will be enrolled for a total of 4 weeks to evaluate the difference in food insecurity, family health measures, and hospital-based quality metrics (including readmission rates and primary care follow up).

ELIGIBILITY:
Inclusion Criteria:

* caregiver and legal guardian of a pediatric patient hospitalized in the acute care units of Brenner Children's Hospital, who have screened positive for food insecurity during the hospitalization.
* lives in the same household as the pediatric patient hospitalized
* lives in Forsyth County, North Carolina
* has a freezer and oven in the household
* does not have family members with food allergies in the household
* willing to accept weekly meal deliveries at home address
* speaks English or Spanish

Exclusion Criteria:

* subjects who do not have the capacity to give legally effective consent
* planning to leave Forsyth County, North Carolina within 6 months of enrollment date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Caregivers Asked to Take Part in Study | Month 4
  Number of caregivers of pediatric inpatients asked to take part in the study.
Number of Caregivers Consented | Month 4
  Number of caregivers of pediatric inpatients who consented to take part in the study.
Number of Meals Delivered | Month 4
  Number of meals delivered to participants in the Meal Delivery arm.
Number of Gift Cards Delivered | Month 4
  Number of gift cards delivered to participants in the Grocery Gift Card arm.
Number of Post-Intervention Surveys Completed | Month 4
  Number of caregivers who completed the post-intervention satisfaction surveys upon study completion.

OTHER OUTCOMES:
Rate of Readmission | Month 4
  Number of caregivers with a child readmitted within 30 days after hospital discharge
Rate of Primary Care Follow Up | Month 4
  Number of caregivers with a child who received primary care follow up after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Leila DeWitt, DO, MA, Principal Investigator — Brenner Children's Hospital
Locations (1):
- Brenner Children's Hospital, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share individual participant data that underlie the results reported after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available immediately after publication with no end date.
Access Criteria: Data will be shared with anyone who wishes to access the data for any purpose. Proposals should be directed to study PI. Data requestors will need to sign a data access agreement.